CLINICAL TRIAL: NCT00155714
Title: Clinical Efficacy of Type-5 Phosphodiesterase Inhibitors (Sildenafil and Vadenafil) in Primary and Secondary Pulmonary Hypertension
Brief Title: Efficacy of Type-5 Phosphodiesterase Inhibitors in Primary and Secondary Pulmonary Hypertension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We can't obtained the test drug (Vadenafil) from Bayer. They decided not to carry out this trail in Taiwan. Therefore this trail has never been started.
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9100017321
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-01

CONDITIONS: Primary and Secondary Pulmonary Hypertension
Keywords: pulmonary arterial hypertension; type-5 phosphodiesterase Inhibitors; Sildenafil
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: type-5 phosphodiesterase Inhibitor (Sildenafil)

SUMMARY:
The aim of this trial is to evaluate the efficacy of type-5 phosphodiesterase inhibitors (sildenafil) in primary and secondary pulmonary hypertension

DETAILED DESCRIPTION:
Patients with primary and secondary pulmonary hypertension will be recruited and admitted to the ICUs of the National Taiwan University Hospital. Each patient will undergo Swan-Ganz catheterization and hemodynamic monitoring during administration of sildenafil. Efficacy of inhaled NO and Iloprost will also be compared.

ELIGIBILITY:
Inclusion Criteria:Patients with primary and secondary pulmonary arterial hypertension

-

Exclusion Criteria:Unstable patients or patients with allergy to sildenafil

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2002-11; Study Completion 2005-05 (Estimated)

PRIMARY OUTCOMES:
mean pulmonary artery pressure
6 min walking distance
WHO functional status
PaO2

SECONDARY OUTCOMES:
cardiac output
VO2max

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Hung Kuo, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Ping-Hung Kuo, Taipei, Taiwan